CLINICAL TRIAL: NCT02104739
Title: Comparative Effects of Antidiabetic Medications on Postprandial Hyperlipidemia, Free Fatty Acid Signaling, and Endothelial Dysfunction in Individuals With Prediabetes
Brief Title: Effects of Antidiabetic Medications on the Postprandial State in Prediabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: The Center for Clinical and Translational Sciences (CCTS) Clinical Research Unit at The University of Texas Health Science Center at Houston (Other)
Responsible Party: Principal Investigator, Absalon D Gutierrez, Assistant Professor of Medicine, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-13-0791
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Prediabetes; Obesity
Keywords: prediabetes; diabetes mellitus type 2; exenatide; saxagliptin; exenatide ER
MeSH Terms: conditions — Prediabetic State; Obesity; Diabetes Mellitus, Type 2 | interventions — Exenatide; saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo pills and placebo injections provided
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (12):
- Exenatide, then Saxagliptin, then Placebo (Experimental): Exenatide Single subcutaneous injection (10 mcg); Saxagliptin Single dose orally (5 mg); Placebo tablets and Placebo (normal saline) injections
  Interventions: Drug: Exenatide; Drug: Saxagliptin; Other: Placebo
- Exenatide, then Placebo, then Saxagliptin (Experimental): Exenatide Single subcutaneous injection (10 mcg); Saxagliptin Single dose orally (5 mg); Placebo tablets and Placebo (normal saline) injections
  Interventions: Drug: Exenatide; Drug: Saxagliptin; Other: Placebo
- Saxagliptin, then Exenatide, then Placebo (Placebo Comparator): Exenatide Single subcutaneous injection (10 mcg); Saxagliptin Single dose orally (5 mg); Placebo tablets and Placebo (normal saline) injections
  Interventions: Drug: Exenatide; Drug: Saxagliptin; Other: Placebo
- Saxagliptin, then Placebo, then Exenatide (Experimental): Exenatide Single subcutaneous injection (10 mcg); Saxagliptin Single dose orally (5 mg); Placebo tablets and Placebo (normal saline) injections
  Interventions: Drug: Exenatide; Drug: Saxagliptin; Other: Placebo
- Placebo, then Exenatide, then Saxagliptin (Experimental): Exenatide Single subcutaneous injection (10 mcg); Saxagliptin Single dose orally (5 mg); Placebo tablets and Placebo (normal saline) injections
  Interventions: Drug: Exenatide; Drug: Saxagliptin; Other: Placebo
- Placebo, then Saxagliptin, then Exenatide (Experimental): Exenatide Single subcutaneous injection (10 mcg); Saxagliptin Single dose orally (5 mg); Placebo tablets and Placebo (normal saline) injections
  Interventions: Drug: Exenatide; Drug: Saxagliptin; Other: Placebo
- Exenatide, then Saxagliptin, then Placebo, then Exenatide ER (Experimental): Exenatide Single subcutaneous injection (10 mcg); Saxagliptin Single dose orally (5 mg); Placebo tablet and Placebo (normal saline) injection; Subcutaneous injection (2mg) weekly for 6 weeks
  Interventions: Drug: Exenatide; Drug: Saxagliptin; Drug: Exenatide extended-release (ER); Other: Placebo
- Exenatide, then Placebo, then Saxagliptin, then Exenatide ER (Experimental): Exenatide Single subcutaneous injection (10 mcg); Saxagliptin Single dose orally (5 mg); Placebo tablet and Placebo (normal saline) injection; Subcutaneous injection (2mg) weekly for 6 weeks
  Interventions: Drug: Exenatide; Drug: Saxagliptin; Drug: Exenatide extended-release (ER); Other: Placebo
- Saxagliptin, then Exenatide, then Placebo, then Exenatide ER (Experimental): Exenatide Single subcutaneous injection (10 mcg); Saxagliptin Single dose orally (5 mg); Placebo tablet and Placebo (normal saline) injection; Subcutaneous injection (2mg) weekly for 6 weeks
  Interventions: Drug: Exenatide; Drug: Saxagliptin; Drug: Exenatide extended-release (ER); Other: Placebo
- Saxagliptin, then Placebo, then Exenatide, then Exenatide ER (Experimental): Exenatide Single subcutaneous injection (10 mcg); Saxagliptin Single dose orally (5 mg); Placebo tablet and Placebo (normal saline) injection; Subcutaneous injection (2mg) weekly for 6 weeks
  Interventions: Drug: Exenatide; Drug: Saxagliptin; Drug: Exenatide extended-release (ER); Other: Placebo
- Placebo, then Exenatide, then Saxagliptin, then Exenatide ER (Experimental): Exenatide Single subcutaneous injection (10 mcg); Saxagliptin Single dose orally (5 mg); Placebo tablet and Placebo (normal saline) injection; Subcutaneous injection (2mg) weekly for 6 weeks
  Interventions: Drug: Exenatide; Drug: Saxagliptin; Drug: Exenatide extended-release (ER); Other: Placebo
- Placebo, then Saxagliptin, then Exenatide, then Exenatide ER (Experimental): Exenatide Single subcutaneous injection (10 mcg); Saxagliptin Single dose orally (5 mg); Placebo tablet and Placebo (normal saline) injection; Subcutaneous injection (2mg) weekly for 6 weeks
  Interventions: Drug: Exenatide; Drug: Saxagliptin; Drug: Exenatide extended-release (ER); Other: Placebo

INTERVENTIONS:
Drug: Exenatide — Single subcutaneous injection (10 mcg)
  Other Names: Byetta
Drug: Saxagliptin — Single dose orally (5 mg)
  Other Names: Onglyza
Drug: Exenatide extended-release (ER) — Subcutaneous injection (2mg) weekly for 6 weeks
  Other Names: Bydureon
  Arms: Exenatide, then Placebo, then Saxagliptin, then Exenatide ER; Exenatide, then Saxagliptin, then Placebo, then Exenatide ER; Placebo, then Exenatide, then Saxagliptin, then Exenatide ER; Placebo, then Saxagliptin, then Exenatide, then Exenatide ER; Saxagliptin, then Exenatide, then Placebo, then Exenatide ER; Saxagliptin, then Placebo, then Exenatide, then Exenatide ER
Other: Placebo — Placebo tablets and Placebo (normal saline) injections

SUMMARY:
This project addresses cardiovascular disease risk in patients with prediabetes. Levels of lipids after eating a meal ("postprandial lipids") are strong independent predictors of cardiovascular risk. Newer anti-diabetic agents - exenatide and saxagliptin - impact lipid metabolism. These medications will be studied for their effect in reducing both postprandial lipid levels and arterial dysfunction.

DETAILED DESCRIPTION:
It is a paradox that medical efforts to control blood glucose in type 2 diabetes mellitus have not decreased the risk of cardiovascular disease. Postprandial lipid concentrations are a strong predictor of cardiovascular risk, independent of traditional cardiovascular risk factors. The new classes of antidiabetic medications - GLP-1 agonists and DPP-IV inhibitors - affect lipid as well as glucose metabolism. This study will investigate the efficacy of these medications in reducing postprandial hyperlipidemia, disrupting the concurrent proinflammatory free fatty acid signaling, and ameliorating endothelial dysfunction in individuals with prediabetes. This will consist of a single center, randomized, crossover, placebo-controlled double-blinded prospective trial involving three study arms representing the aforementioned medications: exenatide (GLP-1 agonist), saxagliptin (DPP-IV inhibitor), and placebo (control arm). Each subject will participate in each of the three arms, which are three separate, daylong outpatient studies. For each study arm, subjects will eat a standardized atherogenic high-fat test lunch. Venous blood draws and measurements of forearm blood flow will be done prior to the meal and periodically during a 6-hour period after the meal. Forearm blood flow measurements will assess for changes in endothelial function. The blood will be analyzed for multiple markers of hyperlipidemia and free fatty acid signaling. After completing the three randomized study visits, subjects are invited to participate in an optional, nonrandomized extension study. For the extension study, subjects will take exenatide ER (extended-release exenatide) weekly for total of six weeks. Then subjects return to eat a standardized atherogenic high-fat test lunch. Venous blood draws and measurements of forearm blood flow will be done prior to the meal and periodically during a 4-hour period after the meal, for the same analyses described before. The results will provide new insights into the anti-inflammatory effects of multiple antidiabetic medications via the mechanisms of postprandial hyperlipidemia, free fatty acid signaling, and endothelial function in prediabetic individuals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Prediabetes - defined as either impaired fasting glucose (fasting glucose of 100-125 mg/dL), impaired glucose tolerance (2-hour postprandial blood glucose of 140-199 mg/dL after 75 gram oral glucose challenge), and/or a hemoglobin A1C ranging from 5.7% to 6.4%
* Subjects are allowed, but not required, to be on statins, ACE-inhibitors, beta-blockers, angiotensin-receptor blockers, thiazide diuretics, and/or loop diuretics at doses that have been stable for at least the last 3 months
* BMI between 30-35 kg/m2 (±1 kg/m2)
* Body weight has been stable (±4-5 pounds) over the prior three months.
* Women of childbearing age must agree to use an acceptable method of pregnancy prevention (barrier methods, abstinence, or surgical sterilization) for the duration of the study
* Patients must have the following laboratory values: Hematocrit ≥ 34 vol% S. creatinine < 1.5 mg/dl in men and 1.4 mg/dl in women AST (SGOT) < 2.5 times ULN, ALT (SGPT) < 2.5 times ULN, alkaline phosphatase< 2.5 times ULN

Exclusion Criteria:

* History of Type 1 or Type 2 diabetes mellitus
* History of diabetic ketoacidosis or hyperosmolar nonketotic coma
* Pregnant or breastfeeding women
* Patients must not be receiving lipid-lowering medications other than statins within the last 3 months
* Patient must not be receiving metformin, DPP-IV inhibitors, GLP-1 agonists, thiazolidinediones, insulin, sulfonylureas, acarbose, SGLT-2 inhibitors, corticosteroids, or immunosuppressive therapy within the last 3 months and cannot take them for the duration of the study. Patient must not be receiving NSAIDS or antioxidant vitamins within the last 1 week, and cannot take them for the duration of the study.
* Patients must not be on hormone replacement therapy.
* Patients with diabetic gastroparesis
* Patients with current tobacco use
* Patients with active malignancy
* Patients with history of urinary bladder cancer
* Patients with dietary restrictions precluding a high-fat meal
* Patients with a history of clinically significant heart disease (NYHA III or IV; more than non- specific ST-T wave changes on the EKG), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation) will not be studied
* Subjects with a history of any serious hypersensitivity reaction to the study medications
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness
* Subjects with known allergic reactions to the study medications or test meal
* Subjects unwilling or unable to provide informed consent
* Subjects determined by the investigator(s) to not be appropriate candidates for the study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Absalaon D Gutierrez, MD, Principal Investigator — University of Texas Health Science Center at Houston, Dept. of Medicine
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Hamidi V, Riggs K, Zhu L, Bermudez Saint Andre K, Westby C, Coverdale S, Dursteler A, Wang H, Miller Iii C, Taegtmeyer H, Gutierrez AD. Acute Exenatide Therapy Attenuates Postprandial Vasodilation in Humans with Prediabetes: A Randomized Controlled Trial. Metab Syndr Relat Disord. 2020 Jun;18(5):225-233. doi: 10.1089/met.2019.0102. Epub 2020 Mar 31. PMID 32228379

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 21 subjects were enrolled. 20 were randomized, and these 20 participated in each of three arms (the exenatide, saxagliptin, and placebo arms), with the order of receipt being randomized. There was an extension phase (that is, the exenatide extended-release (ER) arm) in which 8 of the 21 enrolled participated.
Groups:
- Exenatide, Then Saxagliptin, Then Placebo; Exenatide, Then Placebo, Then Saxagliptin; Saxagliptin, Then Exenatide, Then Placebo; Saxagliptin, Then Placebo, Then Exenatide; Placebo, Then Exenatide, Then Saxagliptin; Placebo, Then Saxagliptin, Then Exenatide; Exenatide Extended-release (Extension Phase): Exenatide arm: Single subcutaneous injection (10 mcg) Saxagliptin arm: Single dose orally (5 mg) Placebo arm: Placebo tablets and Placebo (normal saline) injections Exenatide extended-release (ER) arm: Subcutaneous injection (2mg) weekly for 6 weeks
Period: First Intervention (1 Day)
Arm/Group | Exenatide, Then Saxagliptin, Then Placebo | Exenatide, Then Placebo, Then Saxagliptin | Saxagliptin, Then Exenatide, Then Placebo | Saxagliptin, Then Placebo, Then Exenatide | Placebo, Then Exenatide, Then Saxagliptin | Placebo, Then Saxagliptin, Then Exenatide | Exenatide Extended-release (Extension Phase)
Started | 2 | 5 | 2 | 8 | 0 | 3 | 0
Completed | 2 | 4 | 2 | 7 | 0 | 3 | 0
Not Completed | 0 | 1 | 0 | 1 | 0 | 0 | 0
Period: Washout (Min of 10 and Max of 107 Days)
Arm/Group | Exenatide, Then Saxagliptin, Then Placebo | Exenatide, Then Placebo, Then Saxagliptin | Saxagliptin, Then Exenatide, Then Placebo | Saxagliptin, Then Placebo, Then Exenatide | Placebo, Then Exenatide, Then Saxagliptin | Placebo, Then Saxagliptin, Then Exenatide | Exenatide Extended-release (Extension Phase)
Started | 1 | 4 | 2 | 7 | 0 | 2 | 0
Completed | 1 | 4 | 2 | 7 | 0 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Exenatide, Then Saxagliptin, Then Placebo | Exenatide, Then Placebo, Then Saxagliptin | Saxagliptin, Then Exenatide, Then Placebo | Saxagliptin, Then Placebo, Then Exenatide | Placebo, Then Exenatide, Then Saxagliptin | Placebo, Then Saxagliptin, Then Exenatide | Exenatide Extended-release (Extension Phase)
Started | 1 | 4 | 2 | 7 | 0 | 2 | 0
Completed | 1 | 4 | 2 | 7 | 0 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (Min of 10 and Max of 107 Days)
Arm/Group | Exenatide, Then Saxagliptin, Then Placebo | Exenatide, Then Placebo, Then Saxagliptin | Saxagliptin, Then Exenatide, Then Placebo | Saxagliptin, Then Placebo, Then Exenatide | Placebo, Then Exenatide, Then Saxagliptin | Placebo, Then Saxagliptin, Then Exenatide | Exenatide Extended-release (Extension Phase)
Started | 1 | 4 | 2 | 7 | 0 | 2 | 0
Completed | 1 | 4 | 2 | 7 | 0 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | Exenatide, Then Saxagliptin, Then Placebo | Exenatide, Then Placebo, Then Saxagliptin | Saxagliptin, Then Exenatide, Then Placebo | Saxagliptin, Then Placebo, Then Exenatide | Placebo, Then Exenatide, Then Saxagliptin | Placebo, Then Saxagliptin, Then Exenatide | Exenatide Extended-release (Extension Phase)
Started | 1 | 4 | 2 | 7 | 0 | 2 | 0
Completed | 1 | 4 | 2 | 7 | 0 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (Min of 10 and Max of 323 Days)
Arm/Group | Exenatide, Then Saxagliptin, Then Placebo | Exenatide, Then Placebo, Then Saxagliptin | Saxagliptin, Then Exenatide, Then Placebo | Saxagliptin, Then Placebo, Then Exenatide | Placebo, Then Exenatide, Then Saxagliptin | Placebo, Then Saxagliptin, Then Exenatide | Exenatide Extended-release (Extension Phase)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Extension Phase (6 Weeks)
Arm/Group | Exenatide, Then Saxagliptin, Then Placebo | Exenatide, Then Placebo, Then Saxagliptin | Saxagliptin, Then Exenatide, Then Placebo | Saxagliptin, Then Placebo, Then Exenatide | Placebo, Then Exenatide, Then Saxagliptin | Placebo, Then Saxagliptin, Then Exenatide | Exenatide Extended-release (Extension Phase)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: This was a crossover study in which the 21 who were enrolled participated in each of three arms (the exenatide, saxagliptin, and placebo arms). There was an extension phase (that is, the exenatide extended-release (ER) arm) in which 8 of the 21 enrolled participated.
  Exenatide arm: Single subcutaneous injection (10 mcg) Saxagliptin arm: Single dose orally (5 mg) Placebo arm: Placebo tablets and Placebo (normal saline) injections Exenatide extended-release (ER) arm: Subcutaneous injection (2mg) weekly for 6 weeks
Arm/Group | All Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 3
  More than one race | 1
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16
Height [Mean (Standard Deviation); unit: meters] — Population: Height is reported for those who participated in the three main arms of the study (exenatide, saxagliptin, and placebo arms) but not separately reported for the extension study (extended-release exenatide). All those who participated in the extension study also participated in the three main arms of the study.
  meters | 1.7 (0.11)
Weight [Mean (Standard Deviation); unit: kilograms] — Population: Weight is reported for those who participated in the three main arms of the study (exenatide, saxagliptin, and placebo arms) but not separately reported for the extension study (extended-release exenatide). All those who participated in the extension study also participated in the three main arms of the study.
  kilograms | 93.96 (11.98)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared] — Population: BMI is reported for those who participated in the three main arms of the study (exenatide, saxagliptin, and placebo arms) but not separately reported for the extension study (extended-release exenatide). All those who participated in the extension study also participated in the three main arms of the study.
  kilograms per meter squared | 32.53 (1.92)

OUTCOME MEASURES:

1. Primary Outcome: Monocyte NfkB Levels as Detected by Western Blotting
Description: Monocyte NfkB p65 arbitrary units are quantified by densitometric analysis of the Western blots.
Time Frame: baseline
Measure: Mean (Standard Error); unit: NfkB p65 arbitrary units
Arm/Group | Exenatide | Saxagliptin | Placebo | Exenatide Extended-release (ER)
Number analyzed (Participants) | 16 | 16 | 16 | 7
NfkB p65 arbitrary units | 62.79 (4.05) | 72.03 (6.38) | 67.68 (6.38) | 84.19 (6.45)

2. Primary Outcome: Monocyte NfkB Levels as Detected by Western Blotting
Description: Monocyte NfkB p65 arbitrary units are quantified by densitometric analysis of the Western blots.
Time Frame: 2 hours after ingestion of meal
Measure: Mean (Standard Error); unit: NfkB p65 arbitrary units
Arm/Group | Exenatide | Saxagliptin | Placebo | Exenatide Extended-release (ER)
Number analyzed (Participants) | 16 | 16 | 16 | 7
NfkB p65 arbitrary units | 67.39 (6.44) | 68.39 (5.82) | 71.37 (5.82) | 93.47 (5.69)
Statistical Analysis 1: Comparison: Exenatide; Exenatide at baseline and 2 hours after ingestion of meal is compared; Test type: Superiority; p = 0.27, Non-parametric Wilcoxon paired rank sum
Statistical Analysis 2: Comparison: Saxagliptin; Saxagliptin at baseline and 2 hours after ingestion of meal is compared; Test type: Superiority; p = 0.59, Non-parametric Wilcoxon paired rank sum
Statistical Analysis 3: Comparison: Placebo; Placebo at baseline and 2 hours after ingestion of meal is compared; Test type: Superiority; p = 0.51, Non-parametric Wilcoxon paired rank sum
Statistical Analysis 4: Comparison: Exenatide Extended-release (ER); Exenatide extended-release (ER) at baseline and 2 hours after ingestion of meal is compared; Test type: Superiority; p = 0.31, Non-parametric Wilcoxon paired rank sum

3. Secondary Outcome: Triglycerides
Description: triglycerides
Time Frame: baseline
Population: Data for the exenatide extended-release (ER) arm was only collected at baseline and 2 hours.
Measure: Mean (Standard Error); unit: milligrams per deciliter
Arm/Group | Exenatide | Saxagliptin | Placebo | Exenatide Extended-release (ER)
Number analyzed (Participants) | 16 | 16 | 16 | 7
milligrams per deciliter | 108 (11) | 101 (11) | 102 (14) | 106 (14)

4. Secondary Outcome: Triglycerides
Description: triglycerides
Time Frame: 2 hours after ingestion of meal
Population: Data for the exenatide extended-release (ER) arm was only collected at baseline and 2 hours.
Measure: Mean (Standard Error); unit: milligrams per deciliter
Arm/Group | Exenatide | Saxagliptin | Placebo | Exenatide Extended-release (ER)
Number analyzed (Participants) | 16 | 16 | 16 | 7
milligrams per deciliter | 119 (13) | 130 (16) | 163 (19) | 168 (26)
Statistical Analysis 1: Comparison: Exenatide vs Exenatide Extended-release (ER); Test type: Superiority; p = 0.02, ANOVA

5. Secondary Outcome: Triglycerides
Description: triglycerides
Time Frame: 4 hours after ingestion of meal
Population: Data for the exenatide extended-release (ER) arm was only collected at baseline and 2 hours.
Measure: Mean (Standard Error); unit: milligrams per deciliter
Arm/Group | Exenatide | Saxagliptin | Placebo | Exenatide Extended-release (ER)
Number analyzed (Participants) | 16 | 16 | 16 | 0
milligrams per deciliter | 124 (12) | 153 (24) | 206 (24) |

6. Secondary Outcome: Triglycerides
Description: triglycerides
Time Frame: 6 hours after ingestion of meal
Population: Data for the exenatide extended-release (ER) arm was only collected at baseline and 2 hours.
Measure: Mean (Standard Error); unit: milligrams per deciliter
Arm/Group | Exenatide | Saxagliptin | Placebo | Exenatide Extended-release (ER)
Number analyzed (Participants) | 16 | 16 | 16 | 0
milligrams per deciliter | 161 (24) | 179 (27) | 200 (22) |
Statistical Analysis 1: Comparison: Exenatide vs Saxagliptin; The reported p-value compares exenatide and saxagliptin over all time points (2 hours, 4 hours, 6 hours); Test type: Superiority; p < 0.05, ANOVA
Statistical Analysis 2: Comparison: Exenatide vs Placebo; The reported p-value compares exenatide and placebo over all time points (2 hours, 4 hours, 6 hours); Test type: Superiority; p < 0.05, ANOVA

7. Secondary Outcome: Free Fatty Acids
Description: Free Fatty Acids
Time Frame: baseline
Population: Data for the exenatide extended-release (ER) arm was only collected at baseline and 2 hours.
Measure: Mean (Standard Error); unit: millimoles per liter
Arm/Group | Exenatide | Saxagliptin | Placebo | Exenatide Extended-release (ER)
Number analyzed (Participants) | 16 | 16 | 16 | 7
millimoles per liter | 0.45 (0.04) | 0.49 (0.05) | 0.51 (0.04) | 0.65 (0.05)

8. Secondary Outcome: Free Fatty Acids
Description: Free Fatty Acids
Time Frame: 2 hours after meal
Population: Data for the exenatide extended-release (ER) arm was only collected at baseline and 2 hours.
Measure: Mean (Standard Error); unit: millimoles per liter
Arm/Group | Exenatide | Saxagliptin | Placebo | Exenatide Extended-release (ER)
Number analyzed (Participants) | 16 | 16 | 16 | 7
millimoles per liter | 0.35 (0.05) | 0.18 (0.02) | 0.17 (0.01) | 0.19 (0.05)
Statistical Analysis 1: Comparison: Exenatide vs Exenatide Extended-release (ER); Test type: Superiority; p = 0.018, ANOVA

9. Secondary Outcome: Free Fatty Acids
Description: Free Fatty Acids
Time Frame: 4 hours after meal
Population: Data for the exenatide extended-release (ER) arm was only collected at baseline and 2 hours.
Measure: Mean (Standard Error); unit: millimoles per liter
Arm/Group | Exenatide | Saxagliptin | Placebo | Exenatide Extended-release (ER)
Number analyzed (Participants) | 16 | 16 | 16 | 0
millimoles per liter | 0.43 (0.06) | 0.24 (0.02) | 0.23 (0.02) |

10. Secondary Outcome: Free Fatty Acids
Description: Free Fatty Acids
Time Frame: 6 hours after meal
Population: Data for the exenatide extended-release (ER) arm was only collected at baseline and 2 hours.
Measure: Mean (Standard Error); unit: millimoles per liter
Arm/Group | Exenatide | Saxagliptin | Placebo | Exenatide Extended-release (ER)
Number analyzed (Participants) | 16 | 16 | 16 | 0
millimoles per liter | 0.29 (0.06) | 0.31 (0.02) | 0.33 (0.05) |
Statistical Analysis 1: Comparison: Exenatide vs Saxagliptin; The reported p-value compares exenatide and saxagliptin over all time points (2 hours, 4 hours, 6 hours); Test type: Superiority; p < 0.05, ANOVA
Statistical Analysis 2: Comparison: Exenatide vs Placebo; The reported p-value compares exenatide and placebo over all time points (2 hours, 4 hours, 6 hours); Test type: Superiority; p < 0.05, ANOVA

11. Secondary Outcome: Peak Forearm Blood Flow
Description: Peak forearm blood flow via strain gauge venous occlusion plethysmography
Time Frame: baseline
Population: Though 16 completed the exenatide, saxagliptin, and placebo arms, data is only reported for 15 because the study team was unsuccessful in collecting data for the first study patient. Data for the exenatide extended-release (ER) arm was only collected at baseline and 3 hours.
Measure: Mean (Standard Error); unit: mL per minute per 100mL of tissue
Arm/Group | Exenatide | Saxagliptin | Placebo | Exenatide Extended-release (ER)
Number analyzed (Participants) | 15 | 15 | 15 | 7
mL per minute per 100mL of tissue | 12.65 (1.17) | 12.79 (1.47) | 12.18 (1.17) | 16.18 (1.25)

12. Secondary Outcome: Peak Forearm Blood Flow
Description: Peak forearm blood flow via strain gauge venous occlusion plethysmography
Time Frame: 3 hours after meal
Population: as for outcome 11
Measure: Mean (Standard Error); unit: mL per minute per 100mL of tissue
Arm/Group | Exenatide | Saxagliptin | Placebo | Exenatide Extended-release (ER)
Number analyzed (Participants) | 15 | 15 | 15 | 7
mL per minute per 100mL of tissue | 13.18 (1.21) | 13.25 (1.04) | 15.11 (1.29) | 16.54 (2.23)
Statistical Analysis 1: Comparison: Exenatide vs Exenatide Extended-release (ER); Test type: Superiority; p = 0.5, ANOVA

13. Secondary Outcome: Peak Forearm Blood Flow
Description: Peak forearm blood flow via strain gauge venous occlusion plethysmography
Time Frame: 6 hours after meal
Population: as for outcome 11
Measure: Mean (Standard Error); unit: mL per minute per 100mL of tissue
Arm/Group | Exenatide | Saxagliptin | Placebo | Exenatide Extended-release (ER)
Number analyzed (Participants) | 15 | 15 | 15 | 0
mL per minute per 100mL of tissue | 14.25 (1.09) | 15.87 (1.81) | 13.45 (0.68) |
Statistical Analysis 1: Comparison: Exenatide vs Saxagliptin; The reported p-value compares exenatide and saxagliptin over all time points (3 hours, 6 hours); Test type: Superiority; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Exenatide vs Placebo; The reported p-value compares exenatide and placebo over all time points (3 hours, 6 hours); Test type: Superiority; p > 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Subjects were followed during the study and for 30 days following the last dose. During the cross-over study, subjects were followed for a min of 53 days to a max of 150 days after taking the 1st dose [(3 days for 3, 1-day study arms) + (20 days to 117 days total for 2 washout periods) + 30 = 53 days]. (Washout was at least 20 days but could be 117 days since the cross-over study could span 120 days.) During the extension study, subjects were followed for 72 days after taking the 1st dose.
Arm/Group | Exenatide | Saxagliptin | Placebo | Exenatide Extended-release (ER)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/7
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/7

LIMITATIONS AND CAVEATS:
Lower than expected sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-18): https://cdn.clinicaltrials.gov/large-docs/39/NCT02104739/Prot_SAP_000.pdf